CLINICAL TRIAL: NCT01216735
Title: Effect of an Inhaled Glucocorticosteroid (ICS) on Endothelial Dysfunction in Cigarette Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 20070896; GSK 11340 (Other: Sponsor)
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-05

CONDITIONS: Tobacco Abuse Smoke
Keywords: smokers; inhaled corticosteroids; brachial flow; airway blood flow; albuterol; spirometry; endothelial dysfunction
MeSH Terms: interventions — Fluticasone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- smokers, Fluticasone first, then Placebo (Active Comparator): The current smokers will be given a 3-week treatment course of inhaled fluticasone (220 ug fluticasone twice a day administered as a MDI) . The subjects and the investigators will be blinded to the random choice of inhaler.
  Interventions: Drug: Fluticasone; Drug: Placebo
- smokers Placebo first, then Fluticasone (Placebo Comparator): The current smokers will be given a 3-week treatment course of inhaled placebo MDI. The subjects and the investigators will be blinded to the random choice of inhaler.
  Interventions: Drug: Fluticasone; Drug: Placebo
- health non-smokers (No Intervention): The healthy non-smokers will have only visit 1 and no intervention.

INTERVENTIONS:
Drug: Fluticasone — 220 ug twice a day for 3 weeks
  Other Names: flovent
  Arms: smokers Placebo first, then Fluticasone; smokers, Fluticasone first, then Placebo
Drug: Placebo — Placebo for 3 weeks
  Other Names: sugar pill
  Arms: smokers Placebo first, then Fluticasone; smokers, Fluticasone first, then Placebo

SUMMARY:
The hypothesis underlying the proposed study is that the blunted endothelium-dependent vasodilation seen in the airway of current smokers is also present in the brachial artery, and that the same inhaled corticosteroid (ICS) treatment regime that reversed endothelial function in the airway of current smokers will also restore endothelium-dependent relaxation in the brachial artery. Non-smokers will be used as controls and will not receive any intervention or treatment.

DETAILED DESCRIPTION:
Cigarette smoking can lead to systemic endothelial dysfunction. Since the airway circulation is exposed to a high concentration of cigarette smoke constituents, we reasoned that airway vascular endothelial dysfunction could be present in healthy smokers without systemic endothelial dysfunction.

The purpose of this study was to compare airway and systemic endothelial function and measure markers of systemic inflammation in lung-healthy current smokers. Since endothelial dysfunction in smokers has been related to systemic inflammation, we also investigated its response to an inhaled glucocorticosteroid (ICS).

Vascular endothelial function was assessed in the airway by the airway blood-flow (Qaw) response to inhaled albuterol (ΔQaw) and in the extrapulmonary circulation by brachial arterial flow-mediated vasodilation (FMD). Venous blood was collected for C-reactive protein and IL-6.

Qaw was measured with a noninvasive inhaled soluble gas uptake technique. The uptake of the gas from the anatomical deadspace reflecting airways perfused by the airway circulation was quantitated.

Qaw was express as μL/min normalized for anatomical deadspace: μL/min/mL.

ELIGIBILITY:
Inclusion Criteria:

For both healthy non-smokers and healthy current smokers:

normal spirometry Healthy current smokers: history of >10 pack-year smoking

Exclusion Criteria:

Women of childbearing potential who do not use accepted birth control measures; pregnant and breast feeding women. Cardiovascular disease and/or use of cardiovascular medications. Subjects with known beta-adrenergic agonist or nitroglycerin intolerance. A physician diagnosis of chronic airway disease (asthma, COPD, bronchiectasis, cystic fibrosis).

Acute respiratory infection within four weeks prior to the study. Use of any airway medication. FEV1 < 80% of predicted and FEV1/FVC < 0.7. A body mass index > 30.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- Human Research Laboratory - University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Mendes ES, Campos MA, Wanner A. Airway blood flow reactivity in healthy smokers and in ex-smokers with or without COPD. Chest. 2006 Apr;129(4):893-8. doi: 10.1378/chest.129.4.893. PMID 16608935
- [Background] Mendes ES, Horvath G, Rebolledo P, Monzon ME, Casalino-Matsuda SM, Wanner A. Effect of an inhaled glucocorticoid on endothelial function in healthy smokers. J Appl Physiol (1985). 2008 Jul;105(1):54-7. doi: 10.1152/japplphysiol.90334.2008. Epub 2008 May 8. PMID 18467553
- [Background] Wanner A, Campos MA, Mendes E. Airway blood flow reactivity in smokers. Pulm Pharmacol Ther. 2007;20(2):126-9. doi: 10.1016/j.pupt.2005.12.004. Epub 2006 Jan 18. PMID 16414297

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 Non-smokers were enrolled to provide baseline measures and did not receive any intervention or treatment
Groups:
- Fluticasone First, Then Placebo; Placebo First, Then Fluticasone: The current smokers will be given a 3-week treatment course of inhaled fluticasone (220 ug fluticasone twice a day administered as a MDI) or placebo. The subjects and the investigators will be blinded to the random choice of inhaler.
  Fluticasone: 220 ug twice a day administered as a metered dose inhaled (MDI) or matching placebo
Period: First Intervention (3 Weeks)
Arm/Group | Fluticasone First, Then Placebo | Placebo First, Then Fluticasone
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Washout (3 Weeks)
Arm/Group | Fluticasone First, Then Placebo | Placebo First, Then Fluticasone
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Second Intervention (3 Weeks)
Arm/Group | Fluticasone First, Then Placebo | Placebo First, Then Fluticasone
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 32 participants were enrolled divided in two groups smokers and controls
Groups:
- Smokers: The current smokers will be given a 3-week treatment course of inhaled fluticasone (220 ug fluticasone twice a day administered as a MDI). The subjects and the investigators will be blinded to the random choice of inhaler.
  Fluticasone: 220 ug twice a day administered as a metered dose inhaled (MDI)
- Non-smokers: this group served as controls for baseline data. No intervention or treatment were assigned to this group.
- Total: Total of all reporting groups
Arm/Group | Smokers | Non-smokers | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Full Range); unit: years]
  age | 44 [36 to 58] | 38 [32 to 54] | 42 [32 to 58]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 17 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 15 | 17 | 32
Airway blood flow (Qaw) [Mean (Standard Deviation); unit: um/ml/ul] | 50.3 (3.7) | 46.2 (3.5) | 48.2 (3.4)

OUTCOME MEASURES:

1. Primary Outcome: Albuterol Induced Change in Qaw Before and After Fluticasone or Placebo
Description: Airway Blood flow (Qaw) will be measured before and 15 minutes after albuterol inhalation (delta Qaw).
Time Frame: 3 weeks treatment period of ICS or placebo
Measure: Mean (Standard Error); unit: % change
Groups:
- Fluticasone: The current smokers will be given a 3-week treatment course of inhaled fluticasone (220 ug fluticasone twice a day administered as a MDI). The subjects and the investigators will be blinded to the random choice of inhaler.
  Fluticasone: 220 ug twice a day administered as a metered dose inhaled (MDI)
- Placebo: The current smokers will be given a 3-week treatment course of inhaled placebo MDI. The subjects and the investigators will be blinded to the random choice of inhaler.
  Placebo: Placebo MDI
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 15 | 15
% change | 40.9 (7.3) | 0.0 (3.2)

2. Secondary Outcome: Flow-mediated Brachial Vasodilation (FMD% Peak Delta)
Description: Flow-mediated vasodilation response in the brachial artery will be measured before and 15 minutes.after albuterol inhalation
Time Frame: 3 weeks of treatment
Measure: Mean (Standard Error); unit: % change
Arm/Group | Fluticasone | Placebo
Number analyzed (Participants) | 15 | 15
% change | 3.9 (0.6) | 4.8 (0.6)

ADVERSE EVENTS:
Time Frame: The AEs were collected during the duration of the study.
Groups:
- Fluticasone: The current smokers will be given a 3-week treatment course of inhaled fluticasone (220 ug fluticasone twice a day administered as a MDI). The subjects and the investigators will be blinded to the random choice of inhaler.
  Fluticasone: 220 ug twice a day for 3 weeks
  Placebo: Placebo for 3 weeks
- Placebo: The current smokers will be given a 3-week treatment course of inhaled placebo MDI. The subjects and the investigators will be blinded to the random choice of inhaler.
  Fluticasone: 220 ug twice a day for 3 weeks
  Placebo: Placebo for 3 weeks
Arm/Group | Fluticasone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes